CLINICAL TRIAL: NCT01929109
Title: Pharmacokinetics of LY2409021 Following Administration to Subjects With Varying Degrees of Renal Function
Brief Title: A Study of LY2409021 in Participants With Different Levels of Kidney Function
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 14578; I1R-MC-GLBT (Other: Eli Lilly and Company)
Record Dates: First submitted 2013-08-22; First posted 2013-08-27 (Estimated); Results first posted 2018-10-29 (Actual); Last update posted 2018-10-29 (Actual); Status verified 2018-03

CONDITIONS: Kidney Failure, Chronic; Renal Insufficiency, Chronic
MeSH Terms: conditions — Kidney Failure, Chronic; Renal Insufficiency, Chronic | interventions — adomeglivant

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (5):
- LY2409021 Control (Experimental): Healthy participants received a single 80 mg dose of LY2409021 orally on Day 1 of the study.
  Interventions: Drug: LY2409021
- LY2409021 Mild Renal Impairment (Experimental): Participants received a single 80 mg dose of LY2409021 orally on Day 1 of the study.
  Interventions: Drug: LY2409021
- LY2409021 Moderate Renal Impairment (Experimental): Participants received a single 80 mg dose of LY2409021 orally on Day 1 of the study.
  Interventions: Drug: LY2409021
- LY2409021 Severe Renal Impairment (Experimental): Participants received a single 80 mg dose of LY2409021 orally on Day 1 of the study.
  Interventions: Drug: LY2409021
- LY2409021 End Stage Renal Disease (Experimental): Participants received a single 80 mg dose of LY2409021 orally on Day 1 of Period 1 of the study and a single 80 mg dose of LY2409021 orally on Day 1 of Period 2 of the study.
  Interventions: Drug: LY2409021

INTERVENTIONS:
Drug: LY2409021 — Administered orally

SUMMARY:
The purpose of this study was to measure how much of the study drug, LY2409021, gets into the blood stream and how long it takes the body to get rid of it when given to participants with different levels of kidney function. There were five study groups. Each participant only enrolled in one group. Participants in groups 1 through 4 were healthy or have mild, moderate, or severe kidney disease. They completed one study period lasting about 29 days. Study group 5 enrolled participants with kidney disease who were on dialysis. They have completed two study periods which together last about 59 days. Screening was required within 21 days prior to the start of the study for all participants.

ELIGIBILITY:
Inclusion Criteria:

Inclusion Criteria for ALL Participants

* Male participants must agree to use a reliable method of birth control in addition to having their partner use another method for the duration of the study and for 3 months after the last dose of LY2409021
* Female participants must not be of child-bearing potential
* Participants have a body mass index (BMI) of 18 to 40 kilogram per meter square (kg/m^2), inclusive, at screening

Additional Inclusion Criteria for Control (Healthy) Participants

- Control participants must have normal renal function, assessed by mean estimated creatinine clearance (CLcr) greater than or equal to (≥)90 milliliter per minute (mL/min) at screening and day before dosing

Additional Inclusion Criteria for Participants with Mild-to-Severe Renal Impairment or End Stage Renal Disease (ESRD)

- Males or females with stable mild-to-severe renal impairment, assessed by estimated CLcr, or with ESRD requiring hemodialysis (or hemodiafiltration) for at least 3 months

Additional Inclusion Criteria for Participants with Type 2 Diabetes Mellitus (T2DM)

- Participants with T2DM that are being treated with diet or exercise alone or receive treatment with insulin

Exclusion Criteria:

Exclusion Criteria for ALL Participants

* Participants that require peritoneal dialysis
* Participants that have a current, functioning, organ transplant
* Participants who show evidence of significant active uncontrolled endocrine or autoimmune abnormalities (for example, thyroid disease, pernicious anemia) as judged by the screening physician
* Participants who had a febrile illness within 3 days prior to screening
* Participants with an abnormality in the 12-lead Electrocardiogram (ECG) that, in the opinion of the investigator, increases the risks associated with participating in the study. [Participants with a QT interval corrected using Fridericia's (QTcF) formula >450 millisecond (msec) or a PR interval >0.22 sec on the screening ECG, or who have risk factors for Torsades de Pointes]
* Participants who show evidence of significant active neuropsychiatric disease
* Participants that are currently using or intend to use potent inhibitors of cytochrome P450 (CYP)3A, which include but are not limited to atazanavir, indinavir, nelfinavir, ritonavir, clarithromycin, itraconazole, ketoconazole, nefazodone, saquinavir, and telithromycin
* Participants who are currently using drugs with a narrow therapeutic index (for example, digoxin,lithium, phenytoin, theophylline, and warfarin)
* Participants that are currently using drugs that are known to prolong the QT interval

Additional Exclusion Criteria for Participants with Mild, Moderate or Severe Renal Impairment or ESRD:

* Participants that have used any drug indicated for medical care of the participant's renal impairment, which is not established in dose and administered for at least 7 days before LY2409021 administration
* Participants with poorly controlled hypertension (systolic blood pressure (BP) less than (>)160, diastolic BP >95 mm Hg) and/or evidence of labile blood pressure including symptomatic postural hypotension
* Participants with hemoglobin <9 grams per deciliter (g/dL) or significant active hematologic disease from causes other than underlying renal disease

Additional Exclusion Criteria for Participants with T2DM:

* Participants who use an oral or injectable antihyperglycemic agent, except for insulin, within 1 month prior to dosing (Day 1)
* Participants who have experienced a ketoacidotic episode (pH <7.3) requiring hospitalization in the last 6 months

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2013-08; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (2):
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Munich, Germany
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Liverpool, United Kingdom

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: This study consisted of 5 groups: Group 1-4 (Normal Renal Function Control, Mild, Moderate and Severe Renal Impairment) and Group 5 [End-stage Renal Disease (ESRD)].
Groups:
- LY2409021 Control: Healthy participants received a single 80 milligram (mg) dose of LY2409021 orally on Day 1 of the study.
- LY2409021 End Stage Renal Disease: Participants received a single 80 mg dose of LY2409021 orally on Day 1 of Period 1(Dialysis) of the study and a single 80 mg dose of LY2409021 orally on Day 1 of Period 2 (Non Dialysis) of the study.
Period: Period 1 (All Groups)
Arm/Group | LY2409021 Control | LY2409021 Mild Renal Impairment | LY2409021 Moderate Renal Impairment | LY2409021 Severe Renal Impairment | LY2409021 End Stage Renal Disease
Started | 14 | 8 | 9 | 8 | 8
Completed | 14 | 8 | 8 | 8 | 8
Not Completed | 0 | 0 | 1 | 0 | 0
Not completed — Deviation from protocol | 0 | 0 | 1 | 0 | 0
Period: Period 2 (End Stage Renal Disease Only)
Arm/Group | LY2409021 Control | LY2409021 Mild Renal Impairment | LY2409021 Moderate Renal Impairment | LY2409021 Severe Renal Impairment | LY2409021 End Stage Renal Disease
Started | 0 | 0 | 0 | 0 | 8
Completed | 0 | 0 | 0 | 0 | 8
Not Completed | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | LY2409021 Control | LY2409021 Mild Renal Impairment | LY2409021 Moderate Renal Impairment | LY2409021 Severe Renal Impairment | LY2409021 End Stage Renal Disease | Total
Number analyzed (Participants) | 14 | 8 | 8 | 8 | 8 | 46
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.9 (13.0) | 59.8 (9.1) | 68.6 (6.3) | 63.6 (8.4) | 52.0 (12.0) | 59.2 (11.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 4 | 3 | 1 | 2 | 16
  Male | 8 | 4 | 5 | 7 | 6 | 30
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 1 | 1
  White | 14 | 8 | 8 | 8 | 7 | 45
  More than one race | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0
Type 2 Diabetes Mellitus (T2DM) status [Count of Participants; unit: Participants]
  Yes | 0 | 1 | 0 | 0 | 0 | 1
  No | 14 | 7 | 8 | 8 | 8 | 45
Creatinine clearance (CLcr) [Mean (Standard Deviation); unit: mL/min] — Calculated using the mean of screening and Day -1 values for each individual participant.
  mL/min | 112.686 (16.152) | 72.850 (6.512) | 45.844 (10.121) | 21.951 (3.952) | 13.763 (4.159) | 61.149 (40.837)
Estimated Glomerular Filtration Rate (eGRF) [Mean (Standard Deviation); unit: mL/min/1.73m²] — Calculated using Day -1 values for each individual participant.
  mL/min/1.73m² | 91.272 (17.122) | 68.107 (15.876) | 40.448 (12.793) | 17.565 (7.200) | 8.249 (1.918) | 51.147 (35.467)

OUTCOME MEASURES:

1. Primary Outcome: Pharmacokinetics (PK): Maximum Concentration (Cmax) of LY2409021
Time Frame: Predose, 0.5, 1, 2, 4, 6, 7, 8, 9, 10, 12, 24, 48, 72, 96, 144, 192, 264, 336 hours postdose
Population: All participants in Groups 1-4 who received at least 1 dose of study drug and had evaluable PK data, excluding one participant (discontinued for a protocol violation). No efficacy or safety data for this participant are included in results.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanogram per milliliter (ng/mL)
Groups:
- LY2409021 Control: Healthy participants will receive a single 80 mg dose of LY2409021 orally on Day 1 of the study
- LY2409021 Mild Renal Impairment; LY2409021 Moderate Renal Impairment; LY2409021 Severe Renal Impairment: Participants will receive a single 80 mg dose of LY2409021 orally on Day 1 of the study
Arm/Group | LY2409021 Control | LY2409021 Mild Renal Impairment | LY2409021 Moderate Renal Impairment | LY2409021 Severe Renal Impairment
Number analyzed (Participants) | 14 | 8 | 8 | 8
Nanogram per milliliter (ng/mL) | 2460 (32) | 2320 (30) | 2190 (48) | 2080 (25)

2. Primary Outcome: Pharmacokinetics (PK): Area Under the Concentration Curve From Time Zero to Infinity (AUC 0-∞) of LY2409021
Time Frame: Predose, 0.5, 1, 2, 4, 6, 7, 8, 9, 10, 12, 24, 48, 72, 96, 144, 192, 264, 336 hours postdose
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanogram x hour per milliliter(ng•h/mL)
Arm/Group | LY2409021 Control | LY2409021 Mild Renal Impairment | LY2409021 Moderate Renal Impairment | LY2409021 Severe Renal Impairment
Number analyzed (Participants) | 14 | 8 | 8 | 8
Nanogram x hour per milliliter(ng•h/mL) | 181000 (40) | 179000 (40) | 184000 (56) | 188000 (24)

3. Secondary Outcome: Pharmacokinetics (PK): Maximum Concentration (Cmax) of LY2409021 in Participants With End Stage Renal Disease (ESRD) Before and After Dialysis
Time Frame: Period 1 (Dialysis) and Period 2 (Non Dialysis) Predose, 0.5, 1, 2, 4, 6, 7, 8, 9, 10, 12, 24, 48, 72, 96, 144, 192, 264, 336 hours postdose
Population: All participants in Group 5 who received at least 1 dose of study drug and had evaluable PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Groups:
- LY2409021 End Stage Renal Disease (Dialysis): Participants will receive a single 80 mg dose of LY2409021 orally on Day 1 of Period 1 of the study and a single 80 mg dose of LY2409021 orally on Day 1 of Period 1 of the study.
- LY2409021 End Stage Renal Disease (Non-Dialysis): Participants will receive 80 mg dose of LY2409021 orally on Day 1 of Period 2 of the study.
Arm/Group | LY2409021 End Stage Renal Disease (Dialysis) | LY2409021 End Stage Renal Disease (Non-Dialysis)
Number analyzed (Participants) | 8 | 8
ng/mL | 2120 (72) | 2010 (37)

4. Secondary Outcome: Pharmacokinetics (PK): Area Under the Concentration Curve (AUC) (0-∞) of LY2409021 In Participants With ESRD Before and After Dialysis
Time Frame: Period 1 (Dialysis) and Period 2 (Non Dialysis)- Predose, 0.5, 1, 2, 4, 6, 7, 8, 9, 10, 12, 24, 48, 72, 96, 144, 192, 264, 336 hours postdose
Population: All participants in Group 5 who received at least 1 dose of study drug and had evaluable AUC data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng•h/mL
Groups:
- LY2409021 End Stage Renal Disease (Dialysis): Participants received a single 80 mg dose of LY2409021 orally on Day 1 of Period 1 of the study.
- LY2409021 End Stage Renal Disease (Non-Dialysis): Participants received a single 80 mg dose of LY2409021 orally on Day 1 of Period 2 of the study.
Arm/Group | LY2409021 End Stage Renal Disease (Dialysis) | LY2409021 End Stage Renal Disease (Non-Dialysis)
Number analyzed (Participants) | 8 | 8
ng•h/mL | 119000 (51) | 120000 (37)

ADVERSE EVENTS:
Description: One participant discontinued due to a protocol violation. No efficacy or safety data in results for this participant.
Arm/Group | LY2409021 Control | LY2409021 Mild Renal Impairment | LY2409021 Moderate Renal Impairment | LY2409021 Severe Renal Impairment | LY2409021 End Stage Renal Disease
Serious Adverse Events (participants affected / at risk) | 0/14 | 0/8 | 0/8 | 0/8 | 0/8
Other Adverse Events (participants affected / at risk) | 8/14 | 4/8 | 3/8 | 6/8 | 5/8
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | LY2409021 Control (N=14) | LY2409021 Mild Renal Impairment (N=8) | LY2409021 Moderate Renal Impairment (N=8) | LY2409021 Severe Renal Impairment (N=8) | LY2409021 End Stage Renal Disease (N=8)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Eye irritation (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 1 (2)
Flatulence (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (2) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Fatigue (General disorders) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oedema peripheral (General disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Bronchopneumonia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Oral herpes (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nail injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Procedural site reaction (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Blood phosphorus decreased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Electrocardiogram qt prolonged (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypoglycaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Dysgeusia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Loss of consciousness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)

LIMITATIONS AND CAVEATS:
One participant who received drug was identified as deviating from the protocol due to having Type 1 Diabetes Mellitus (T1DM) and was discontinued and data are not included in Baseline Characteristics, Outcome Measures or AEs.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less